CLINICAL TRIAL: NCT03108716
Title: Hamate Hook Removal, Microscrew Internal Fixation and Plaster Fixation for the Treatment of Hamate Hook Fractures: a Case Series
Brief Title: Hamate Hook Removal, Microscrew Internal Fixation and Plaster Fixation for the Treatment of Hamate Hook Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siping Central People's Hospital (Other)
Responsible Party: Principal Investigator, Zhuang Liu, Principal Investigator, Siping Central People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SipingCPH_001
Record Dates: First submitted 2017-04-05; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Fractures, Bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Intervention Model Description: The investigators collected data of 28 hamate hook fractures patients, who were treated in the Siping Central People's Hospital and had complete follow-up records.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- hamate hook removal (Experimental): The patients were assigned to hamate hook removal(n=13).
  Interventions: Procedure: hamate hook removal
- microscrew internal fixation (Experimental): The patients were assigned to the microscrew internal fixation after open reduction (n=11).
  Interventions: Procedure: microscrew internal fixation
- short-arm tube-type plaster fixation (Experimental): The patients were assigned to the short-arm tube-type plaster fixation (conservative treatment) (n=4).
  Interventions: Other: short-arm tube-type plaster fixation

INTERVENTIONS:
Procedure: hamate hook removal — The patients were assigned to treat with hamate hook removal.
  Arms: hamate hook removal
Procedure: microscrew internal fixation — The patients were assigned to treat with microscrew internal fixation after open reduction.
  Arms: microscrew internal fixation
Other: short-arm tube-type plaster fixation — The patients were assigned to treat with short-arm tube-type plaster fixation (conservative treatment).
  Arms: short-arm tube-type plaster fixation

SUMMARY:
To compare the effects of hamate hook removal, microscrew internal fixation and plaster fixation on fracture healing, work, life, and exercise recovery in patients with hamate hook fractures by retrospective case analysis.

DETAILED DESCRIPTION:
Hamate hook fractures are rare, and mainly occur during sports activities. Its projection is often obscured by other carpal bone in conventional X-ray plain films, so hamate hook fractures are the most easily missed injury in hand surgery. As the incidence of such fractures is too small, it brings some difficulties in the clinical choice of correct and effective treatment. Currently, treatment programs of hamate hook fractures also are not consistent.

ELIGIBILITY:
Inclusion Criteria:

* Hamate hook fractures finally diagnosed by X-ray and CT scan at the wrist position holding a cup and the carpal canal position (appendix 2)
* Unilateral hamate hook fractures
* Irrespective of age and sex

Exclusion Criteria:

* Incomplete follow-up data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Fracture healing | At 6-18 months after surgery
  Fracture healing was assessed using CT images or X-ray films at the wrist position holding a cup.

SECONDARY OUTCOMES:
Time of plaster fixation | At 6-18 months after surgery
  To reflect fracture healing; the shorter the fixation time, the faster the healing

CONTACTS AND LOCATIONS:
Overall Officials: Zhuang Liu, Ph.D, Principal Investigator — Siping Central People's Hospital

IPD SHARING:
Plan to Share IPD: Undecided